CLINICAL TRIAL: NCT02779764
Title: A Phase 3, Long-term Study of Intermittent Oral Dosing of ASP1517 in Hemodialysis Chronic Kidney Disease Patients With Anemia Converted From Erythropoiesis Stimulating Agent Treatment
Brief Title: A Long Term Study of Intermittent Oral Dosing of ASP1517 in Hemodialysis Chronic Kidney Disease Patients With Anemia Converted From Erythropoieses Stimulating Agent (ESA) Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-0312
Record Dates: First submitted 2016-05-19; First posted 2016-05-20 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hemodialysis Patients With Renal Anemia
Keywords: Hemodialysis; ASP1517; Roxadustat; Renal anemia
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASP1517 Group (Experimental): Study drug will be dosed three times weekly and dose adjustments will be made during the study.
  Interventions: Drug: roxadustat

INTERVENTIONS:
Drug: roxadustat — Oral
  Other Names: ASP1517

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ASP1517 in hemodialysis patients with renal anemia whose treatment is converted from an Erythropoieses Stimulating Agent formulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with renal anemia who have been receiving ESA (intravenous treatment) within the doses approved in Japan for more than 8 weeks before the screening assessment
* Mean of the subject's two most recent Hb values during the Screening Period must be ≥10.0 g/dL and ≤12.0 g/dL.
* Either transferrin saturation (TSAT) ≥ 20% or serum ferritin ≥ 100 ng/mL during the screening period
* Female subject must either:

Be of non-childbearing potential:

* post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
* documented surgically sterile Or, if of childbearing potential,
* Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
* And have a negative pregnancy test at Screening
* And, if heterosexually active, agree to consistently use two forms of highly effective birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and continued for 28 days after the final study drug administration.

  * Female subject must agree not to breastfeed starting at Screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Female subject must not donate ova starting at Screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Male subject and their female spouse/partners who are of childbearing potential must be using two forms of highly effective birth control (at least one of which must be a barrier method) starting at Screening and continue throughout the study period, and for 12 weeks after the final study drug administration
  * Male subject must not donate sperm starting at Screening and throughout the study period and, for 12 weeks after the final study drug administration

Exclusion Criteria:

* Concurrent retinal neovascular lesion requiring treatment and macular edema requiring treatment
* Concurrent autoimmune disease with inflammation that could impact erythropoiesis
* History of gastric/intestinal resection considered influential on the absorption of drugs in the gastrointestinal tract (excluding resection of gastric or colon polyps) or concurrent gastro-paresis
* Uncontrolled hypertension
* Concurrent congestive heart failure (NYHA Class III or higher)
* History of hospitalization for treatment of stroke, myocardial infarction, or pulmonary embolism within 12 weeks before the screening assessment
* Positive for hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV) antibody at the screening assessment, or positive for human immunodeficiency virus (HIV) in a past test
* Concurrent other form of anemia than renal anemia
* Having received treatment with protein anabolic hormone, testosterone enanthate, or mepitiostane within 6 weeks before the screening assessment
* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), or total bilirubin that is greater than the criteria, or previous or concurrent another serious liver disease at screening assessment
* Previous or current malignant tumor (no recurrence for at least 5 years is eligible.)
* Having undergone blood transfusion and/or a surgical procedure consider to promote anemia (excluding shunt reconstruction surgery for access to the blood) within 4 weeks before the screening assessment
* Having undergone a kidney transplantation
* Having a previous history of treatment with ASP1517
* History of serious drug allergy including anaphylactic shock
* Participation in another clinical study or post-marketing clinical study (including that of a medical device) within 12 weeks before informed consent acquisition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (Hb) Response Rate from Week 18 to Week 24 | Week 18 to 24
  Hb response defined as average Hb within the target range

SECONDARY OUTCOMES:
Hb Response Rate from Week 46 to Week 52 | Week 46 to 52
Average Hb from Week 18 to Week 24 | Week 18 to Week 24
Average Hb from Week 46 to Week 52 | Week 46 to Week 52
Change from baseline in the average Hb from Week 18 to Week 24 | Baseline and Weeks 18 to 24
Change from baseline in the average Hb from Week 46 to Week 52 | Baseline and Weeks 46 to 52
Proportion of participants with Hb values within the target value in each post-dosing time point | Up to Week 52
Change from baseline in Hb to each post-dosing time point | Baseline and Up to Week 52
Proportion of measurement points with target Hb level from Week 18 to Week 24 | Week 18 to Week 24
Proportion of measurement points with target Hb level from Week 46 to Week 52 | Week 46 to Week 52
Rate of rise in Hb levels (g/dL/week) from week 0 to at the earliest date of week 4, time of discontinuation, or time of dose adjustment | Up to Week 4
Average hematocrit level | Up to Week 52
Average reticulocyte level | Up to Week 52
Average Fe level | Up to Week 52
Average ferritin level | Up to Week 52
Average transferrin level | Up to Week 52
Average total iron binding capacity level | Up to Week 52
Average soluble transferrin receptor level | Up to Week 52
Average transferrin saturation level | Up to Week 52
Average reticulocyte hemoglobin content level | Up to Week 52
Quality of life assessed by SF-36 | Up to Week 52
  SF-36: Medical Outcomes Study 36-Item Short-Form Health Survey
Quality of life assessed by EQ-5D | Up to Week 52
  EQ-5D: EuroQol 5 Dimension
Quality of life assessed by FACT-An | Up to Week 52
  FACT-An: Functional Assessment of Cancer Therapy-Anemia
Number of hospitalizations | Up to Week 52
Safety assessed by incidence of adverse events | Up to Week 52
Number of participants with abnormal Vital signs and/or adverse events related to treatment | Up to Week 52
  Vital signs: blood pressure and pulse rate
Safety assessed by standard 12-lead electrocardiogram | Up to Week 52
Number of participants with abnormal Laboratory values and/or adverse events related to treatment | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (25):
- Japan (25):
  - Site JP00017, Aichi
  - Site JP00005, Fukuoka
  - Site JP00004, Gunma
  - Site JP00006, Gunma
  - Site JP00018, Hokkaido
  - Site JP00019, Hokkaido
  - Site JP00021, Hokkaido
  - Site JP00023, Hyōgo
  - Site JP00008, Ibaraki
  - Site JP00020, Ishikawa
  - Site JP00010, Kumamoto
  - Site JP00022, Kumamoto
  - Site JP00024, Kumamoto
  - Site JP00016, Kyoto
  - Site JP00002, Nagano
  - Site JP00012, Nagano
  - Site JP00015, Nagano
  - Site JP00003, Niigata
  - Site JP00025, Osaka
  - Site JP00007, Saitama
  - Site JP00009, Shizuoka
  - Site JP00014, Tokyo
  - Site JP00013, Tottori
  - Site JP00011, Wakayama
  - Site JP00001, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Hamano T, Yamaguchi Y, Goto K, Mizokawa S, Ito Y, Dellanna F, Barratt J, Akizawa T. Risk Factors for Thromboembolic Events in Patients With Dialysis-Dependent CKD: Pooled Analysis of Phase 3 Roxadustat Trials in Japan. Adv Ther. 2024 Apr;41(4):1526-1552. doi: 10.1007/s12325-023-02727-3. Epub 2024 Feb 16. PMID 38363463
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=358